CLINICAL TRIAL: NCT03796104
Title: Prognostic Impact of Delta-haemolysin Production Deficiency in Staphylococcus Aureus on the Prognosis of Infected Implant Treated by DAIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, clinical research assistant, Hospices Civils de Lyon
Other Study IDs: 18-333
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bone and Joint Infection; Staphylococcus Aureus
Keywords: Bone and Joint Infection; Staphylococcus Aureus; chronic infection
MeSH Terms: conditions — Staphylococcal Infections; Persistent Infection | interventions — delta hemolysin protein, Staphylococcus aureus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deficiency of delta-hemolysine: Implant infected by Staphylococcus aureus with delta-haemolysin Production Deficiency
  Interventions: Other: Delta-haemolysin
- Presence of delta-hemolysine: Implant infected by Staphylococcus aureus with delta-haemolysin Production
  Interventions: Other: Delta-haemolysin

INTERVENTIONS:
Other: Delta-haemolysin — comparison of groups having infection with S. aureus with and without delta-haemolysin Production

SUMMARY:
The aim of this study is to determine if delta-haemolysin production deficiency of Staphylococcus aureus is a marker in favour of chronic infections on implants

ELIGIBILITY:
Inclusion Criteria:

* patients having implant infection due to S. aureus treated by DAIR

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having implant infection due to S. aureus treated by DAIR managed at the Lyon Bone and joint infection reference Center between 2006 and 2018
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of infection with or witout delta-haemolysin in Staphylococcus Aureus | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  patients, profile of the bacterium, medical and chirurgical treatment, rate. comparison between the 2 groups

SECONDARY OUTCOMES:
Rate of Treatment Failure | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin. Analyse of risk factor. Comparison between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: FLORENT VALOUR, Md,PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided